CLINICAL TRIAL: NCT04934891
Title: A Double-Blind, Placebo-Controlled, Dose-Escalation Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of ION547 Administered Subcutaneously to Healthy Subjects
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of ION547
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ION547-CS1
Record Dates: First submitted 2021-06-08; First posted 2021-06-22 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers
Keywords: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ION547 (Experimental): Ascending single multiple doses of ION547 will be administered by SC injection.
  Interventions: Drug: ION547
- Placebo (Placebo Comparator): Ascending single multiple doses of ION547-matching placebo will be administered by SC injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ION547 — ION547 will be administered by SC injection.
  Arms: ION547
Drug: Placebo — ION547-matching placebo will be administered by SC injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single and multiple doses of the antisense inhibitor ION547 administered subcutaneously (SC) in healthy participants.

DETAILED DESCRIPTION:
This is a Phase 1, double-blind, randomized, placebo-controlled, dose escalation study of ION547 in up to 76 participants. Participants will be randomized to receive single and multiple doses of ION547 or placebo SC. The maximum length of participation in the study will be approximately 34 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated) and any authorizations required by local law and be able to comply with all study requirements.
2. Healthy males or females 18 to 65, inclusive, at the time of informed consent.
3. Satisfy the following:

   a. Females: Women of childbearing potential are not allowed to participate in this study.
4. b. Males must be abstinent, surgically sterile (vasectomy with negative semen analysis at Follow-up, or a surgically sterile non-pregnant female partner) or if engaged in sexual relations with a woman of childbearing potential (WOCBP), participant is utilizing a highly effective contraceptive method
5. Body mass index (BMI) ≤ 35 kilograms per square meter (kg/m^2).

Exclusion Criteria:

1. Clinically significant abnormalities in medical history or physical examination.
2. Screening laboratory results as follows, or any other clinically significant (CS) abnormalities in screening laboratory values that would render a participant unsuitable for inclusion:

   1. Urine protein/creatinine (P/C) ratio greater than or equal to (≥) 0.2 milligrams (mg)/mg.
   2. Positive test (including trace) for blood on urinalysis.
   3. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, alkaline phosphatase (ALP), serum creatinine, and blood urea nitrogen (BUN) > upper limit of normal (ULN).
   4. Hemoglobin A1c (HbA1c) > ULN
   5. Platelet count < lower limit of normal (LLN)
   6. aPTT > ULN
   7. INR > 1.4
   8. Evidence of uncorrected hypothyroidism or hyperthyroidism based on thyroid function results at Screening.
3. Uncontrolled hypertension (blood pressure [BP] > 160/100 millimeters of mercury [mmHg]).
4. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
5. Treatment with another investigational drug, biological agent, or device within 1 month of Screening, or 5 half-lives of investigational agent, whichever is longer.
6. Previous treatment with an oligonucleotide (including small interfering ribonucleic acid [siRNA]) within 4 months of screening if single dose received, or within 12 months of screening if multiple doses received. Exclusion does not apply to Covid-19 messenger ribonucleic acid (mRNA) vaccines.
7. History of bleeding diathesis or coagulopathy.
8. Regular use of alcohol within 6 months prior to screening (> 7 drinks/week for females, > 14 drinks/week for males [1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor]), or use of soft drugs (such as marijuana) within 3 months prior to screening, or hard drugs (such as cocaine and phencyclidine [PCP]) within 1 year prior to screening, or positive urine drug screen at Screening.
9. Concomitant medication restrictions: the use of prescription and over-the-counter medications including nonsteroidal anti-inflammatory drugs (with the exception of occasional acetaminophen or ibuprofen) and herbal remedies at Screening and throughout the Study Period.
10. Smoking limitations: more than 10 cigarettes/day at Screening and those with a significant change in smoking habits within 1 month prior to Screening should be excluded.
11. Blood donation of 50 to 499 mL within 30 days of Screening or of > 499 mL within 60 days of Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE) | Up to Day 232
Cmax: Maximum Observed Plasma Concentration of ION547 | Up to Day 232
Tmax: Time Taken to Reach Maximal Plasma Concentration of ION547 | Up to Day 232
AUCt: Area Under the Plasma Concentration-time Curve From Time Zero to Time t for ION547 | Up to Day 232
Urine 0-24 Hour (hr) Excretion of ION547 | Up to 24 hours
Change from Baseline in FXII Antigen Levels | Up to Day 232
Change from Baseline in FXII Activity Levels | Up to Day 232

CONTACTS AND LOCATIONS:
Locations (1):
- BioPharma Services, Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No